CLINICAL TRIAL: NCT02102269
Title: Sonographic Evaluation of the Effect of Shoulder Orthosis on the Subluxation in Stroke Patients
Acronym: SinSbyS&Co
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EC/2013/991
Record Dates: First submitted 2014-03-17; First posted 2014-04-02 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Stroke Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- actimove sling (Active Comparator): standard orthosis: actimove sling
  Interventions: Device: actimove sling
- shoulderlift (Experimental): newly developed orthosis: shoulderlift
  Interventions: Device: shoulderlift
- controle group (No Intervention): no orthosis

INTERVENTIONS:
Device: actimove sling
  Arms: actimove sling
Device: shoulderlift
  Arms: shoulderlift

SUMMARY:
Shoulder pain is frequently reported as a complication among stroke patients. Muscular imbalance disrupts stability of the glenohumeral joint creating a subluxation. Stretching the soft tissue can cause shoulder pain which impedes quality of life, length of stay and rehabilitation outcome. To align the humeral head in the cavitas glenoïdalis a shoulder orthosis is often provided to the patient. Since the use of these orthoses is not always considered positive by the patient nor the therapist the question rises if the investigators can objectify if the subacromial space is reduced when wearing a sling.

Sonography is a valid way to asses subluxation of the shoulder joint by measuring the subacromial space. To objectify if an orthosis can reduce the enlarged subacromial space the investigators will use sonography to measure the distance between acromion and greater tuberosity are between acromion and the humeral head. This distance will be measured with and without the orthosis and also after a period of at least 4 hours of wearing the orthosis. This last measurement might inform us about how long the orthosis can correct the glenohumeral position. To validate the sonographic measurement X-rays will be taken by a sample of the investigators study population to compare with the ultrasound data.

Two different orthoses will be compared. First of all the actimove sling, which is standardly used in the rehabilitation centre where patients will be recruited. This sling can be adapted by the patient itself and is very easy to wear. The disadvantage is that the elbow is continuously flexed, which enlarges the risk on contractures of m. biceps and m. brachioradialis. Also the negative influence on the interpretation of the body scheme and on the quantitative use of the arm can be reasons not to wear this kind of orthosis. The shoulderlift on the other hand is a newly developed orthosis which supports the shoulder joint with the arm extended. This is a more normal position during the daily living and stimulates the use of the paretic arm. An extra adaptation can be adjusted to make it possible to position the arm flexed in order to reduce oedema of the hand if necessary. The control group does not wear any orthosis at all.

Additional the investigators will evaluate passive range of motion of the shoulder, spasticity of the upper limb (modified ashworth scale), active motion of the upper limb (fugl meyer assessment) and trunk stability (Trunk Impairment Scale) at starting point and after a period of 6 weeks wearing the orthosis minimal 6 hours a day.

If possible the investigators will do an evaluation of balance on a moving platform and an evaluation of gait with and without the orthosis after 6 weeks to assess the impact of on balance and gait.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* Patients must be able to sit independently on a chair with arm support during 30 minutes

Exclusion Criteria:

* No shoulder problems prior to stroke
* No severe cognitive problems that make it impossible to understand brief commands;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Acromio - humeral distance | at 9 weeks after admission in the rehabilitation center
Acromio - humeral distance | at 3 weeks after admission in the rehabilitation center

SECONDARY OUTCOMES:
Spasticity | at 9 weeks after admission in the rehabilitation center
  Modified Ashworth Scale
Passive Range of motion | at 9 weeks after admission in the rehabilitation center
  goniometric measurement
Trunk stability | at 9 weeks after admission in the rehabilitation center
  Trunk Impairment Scale
comfort of the upper limb | at 9 weeks after admission in the rehabilitation center
  Pain and comfort questionnaire
Balance | at 9 weeks after admission in the rehabilitation center
Gait characteristics | at 9 weeks after admission in the rehabilitation center
  Measurement: Gait Rite
Spasticity | at 3 weeks after admission in the rehabilitation center
  Modified Ashworth Scale
Passive Range of motion | at 3 weeks after admission in the rehabilitation center
  goniometric measurement
Trunk stability | at 3 weeks after admission in the rehabilitation center
  Trunk Impairment Scale
comfort of the upper limb | at 3 weeks after admission in the rehabilitation center
  Pain and comfort questionnaire
Balance | at 3 weeks after admission in the rehabilitation center
Gait characteristics | at 3 weeks after admission in the rehabilitation center
  Measurement: Gait Rite
Pain of the upper limb | at 3 weeks after admission in the rehabilitation center
  Pain and comfort questionnaire
Pain of the upper limb | at 9 weeks after admission in the rehabilitation center
  Pain and comfort questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Cambier, MD, PhD, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Department of Physical and Rehabilitation Medicine, Ghent
  - Ghent University, Department of Rehabilitation Sciences and Physiotherapy, Ghent